CLINICAL TRIAL: NCT00154700
Title: A Phase II Study of Twice Weekly Paclitaxel, Cisplatin and Weekly 24-Hour Infusion of High-Dose 5-Fluorouracil and Folinic Acid in the Treatment of Recurrent or Metastatic Esophageal Cancer
Brief Title: Twice Weekly TP-HDFL for Recurrent or Metastatic Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 159I9
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-07

CONDITIONS: Esophageal Cancer
Keywords: Combination,Chemotherapy,Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel,Cisplatin,5-Fu,Folic Acid

SUMMARY:
The primary objective of this study is to find out the response rate of twice weekly paclitaxel and cisplatin and weekly HDFL in recurrent or metastatic esophageal carcinoma patients who need palliative Chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to find out the response rate of twice weekly paclitaxel and cisplatin and weekly HDFL in recurrent or metastatic esophageal carcinoma patients who need palliative Chemotherapy. The secondary objectives include overall survival, progression-free survival, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven esophageal squamous cell or adenocarcinoma Recurrence or metastasis Measurable disease (> 1 X 1 cm) by CXR, CT scan or MRI,Age > 18, KPS > 60% , Cre < 1.5mg/dl, AST/ALT < 3.5 X N, Bil < 2.0mg/dl WBC > 4,000/mm3, ANC > 2,000/ mm3, Plt > 100,000/mm3

Exclusion Criteria:

* Prior chemo (except as radiosensitizers)Recurrent, treated esophageal lesion only (except > 2 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-01; Study Completion 2005-07

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Overall survival
Progression-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, M.D., Ph.D., Study Chair — Department of Oncology, National Taiwan University hospital; Ann-Lii Cheng, M.D.,Ph.D, Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan